CLINICAL TRIAL: NCT03867903
Title: BabySparks© App: A Pilot Study of mHealth Adherence to a Developmental Application for Infants After Neonatal Cardiac Surgery
Brief Title: BabySparks Developmental Application Pilot Study
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Lori Erickson, Director Remote Health Solutions, Children's Mercy Hospital Kansas City
Other Study IDs: Study00000385
Record Dates: First submitted 2019-03-01; First posted 2019-03-08 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Development, Child; Adherence, Patient; Congenital Heart Disease
MeSH Terms: conditions — Patient Compliance; Heart Defects, Congenital | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Babysparks Application — mHealth application, BabySparks©, will be implemented for infant and toddler developmental activities through 24 months of age. (Currently, BabySparks is only designed to work on the developmental milestones through 24 months of age, and therefore the use of the application will no longer be applicable to the patient after reaching a developmental age of 24 months. If the subject has not reached a developmental age of 24 months at the time he/she is chronologically 24 months, the subject/family will be able to continue to utilize the application for a maximum of 24 months from the time they began to use the application or until reaching a study endpoint of reaching 24 months developmentally or death, whichever the infant reaches first.)
Other: pre and post-test Redcap Survey — Prior to starting the use of the application, parents will be given a REDCap survey to complete to determine their current awareness and interventions being implemented with their child related to reaching developmental milestones. Data entered into application by the subject's caregivers will be stored by BabySparks.After completion of the use of the application (subject reaches a study endpoint), the caregivers will be asked to complete a REDCap survey asking them about their experience with the application.

SUMMARY:
A single site, cross-sectional, pilot study of a mHealth application. Primary Objective This purpose of this pilot study is to evaluate mHealth adherence to a developmental application, Babysparks©, by parents of infants with complex congenital cardiac disease and single ventricle heart disease.

Secondary Objective(s) -To determine the demographic and infant characteristics that correlate with mHealth adherence.

-The rate of developmental progress of milestones while using the application will also be compared between infants with single ventricle cardiac disease and bi-ventricular cardiac disease.

Research Intervention(s)/ Investigational Agent(s) Babysparks© developmental application is the main intervention with evaluation on feasibility of the mHealth application in a pediatric cardiology population.

Study participants will be parents of infants with single ventricle and bi-ventricular complex congenital heart disease who underwent cardiac surgery in the first six weeks of life and are currently less than 18 months of age.

Study Population There are approximately 150 new patients a year who have undergone cardiac surgery, with an additional 150 who are 18 months of age or less.

Sample Size A maximum of 400 families/year Study Duration for Individual Participants Study participants will be monitored for a minimum of 6 months with the use of the BabySparks© App; to a maximum of 24 months of use of the app or when the child reaches a developmental age of 24 months, whichever occurs first.

Study Specific Abbreviations/ Definitions mHealth : mobile health CHD: Congenital heart disease

DETAILED DESCRIPTION:
Study design. A single site, cross-sectional, pilot study, with a pre/post-test design will be used to evaluate the mHealth adherence and the parental feedback after using this application. Additional feasibility measures of the application will be evaluated through the engagement and use of the application, use of the mHealth data back to the research team, and frequency of the parents implementing app-suggested activities, and the infants' ability to complete these developmental activities during use of the application.

Theoretical Framework. Pediatric self-management theoretical framework follows infants to adolescents on a dynamic continuum with frequent modifiable and non-modifiable factors, processes, and behaviors that may affect adherence and outcomes. The factors may come from individual non-modifiable congenital heart disease, family factors, community support, and the health care system where the infant has their care. The interplay between parental stress and adherence to developmental interventions are highlighted in this theoretical framework, and allows for an underpinning framework for this study. Previous work with parental caregiving and motivation has included a theoretical model of the attachment-parenting theory which also supports this study to encourage interactive behaviors and developmental interventions.

Research Procedures: The mHealth application will be downloaded by parents onto up to 5 devices of their choosing with a primary email address as the linking account.

The parents will be sent a REDCap survey prior to starting the use of the application to determine their current awareness and interventions being implemented with their child related to reaching developmental milestones, and a second survey will be sent to the family at the end of study period to get their feedback on the mHealth application.

Data to be collected from the Electronic medical record (Stored in REDcap form), none of these are going to be stored in an identifiable manner: Cardiac diagnosis, Prenatal diagnosis, Cardiac surgery, Major genetic diagnosis, Major non-cardiac diagnosis, Age in days of cardiac surgery, Length of neonatal hospitalization (Days), Used the app prior to discharge, Age in days when parent started using the application, Total number of days in the hospital the first year of life, Total number of ICU days in the first year of life, Primary parent age, Primary parent gender, Primary parent education level, Number of other siblings, Route of feeds at discharge, Distance from the hospital at home

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be infants (and their parents) who have undergone cardiac surgery at Children's Mercy Kansas City in the first six weeks of life and are currently less than 18 months of age at the time of being approached for participation in this study.

Exclusion Criteria:

* • Families without access to a personal device for download (no devices will be provided)

  * Children who are deceased prior to the family being approached for study participation
  * Neonates that are considered non-viable, or have the potential to be non-viable
  * Spanish-only speaking families

Exclude special populations:

• Wards of the state

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with single ventricle cardiac disease are also known to have more complex hospitalizations and need for gastrostomy feeding tubes as compared to infants with bi-ventricular cardiac disease. The need for gastrostomy feeding is associated with a higher risk of cognitive, language, and motor delays in toddler age children with cardiac disease with Post-acute care interventions for physical and occupational therapy like "tummy time" are recommended for infants, but there is a lack of specific guidelines or recommendations in pediatric cardiac programs related to the use of mHealth interventions performed by parents after their discharge to home.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Acceptability | At end of 6 months Redcap Survey
  satisfaction assessed through the end point survey
Adoption | Date of Download of the application to the parent phone assessed 1 month
  through uptake of application onto the phone
initial implementation | First date used after download onto parent phone assessed in 1 month
  first date used after download
Utilization | 6 months after study enrollment
  Frequency of use after download
Appropriateness | at end of study Redcap Survey ( 6 months after study enrollment)
  Parental Feedback from endpoint survey on appropriate developmental questions and interventions for their child

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, MSN, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modi AC, Pai AL, Hommel KA, Hood KK, Cortina S, Hilliard ME, Guilfoyle SM, Gray WN, Drotar D. Pediatric self-management: a framework for research, practice, and policy. Pediatrics. 2012 Feb;129(2):e473-85. doi: 10.1542/peds.2011-1635. Epub 2012 Jan 4. PMID 22218838
- [Background] McKechnie AC, Rogstad J, Martin KM, Pridham KF. An exploration of co-parenting in the context of caring for a child prenatally diagnosed and born with a complex health condition. J Adv Nurs. 2018 Feb;74(2):350-363. doi: 10.1111/jan.13415. Epub 2017 Oct 4. PMID 28792608
- [Background] McWilliams A, Reeves K, Shade L, Burton E, Tapp H, Courtlandt C, Gunter A, Dulin MF. Patient and Family Engagement in the Design of a Mobile Health Solution for Pediatric Asthma: Development and Feasibility Study. JMIR Mhealth Uhealth. 2018 Mar 22;6(3):e68. doi: 10.2196/mhealth.8849. PMID 29567637